CLINICAL TRIAL: NCT04080908
Title: Open Label Single Arm Pilot Study to Assess Feasibility and Safety of Iron Repletion With Feraheme in Iron Deficient Patients With Durable Ventricular Assist Device Support
Brief Title: Study to Assess Feasibility and Safety of Iron Repletion With Feraheme in Iron Deficient Patients With Durable Ventricular Assist Device Support
Acronym: AMAGFeraheme
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to meet enrollment goals.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-00866
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Results first posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ferumoxytol injection treatment (Experimental)
  Interventions: Drug: Ferumoxytol injection

INTERVENTIONS:
Drug: Ferumoxytol injection — Two doses of ferumoxytol injection will be administered intravenously 3-8 days apart.

SUMMARY:
Ferumoxytol injection (Feraheme®) is a parenteral form of iron supplementation that is FDA-approved for treatment of iron deficiency anemia. Ferumoxytol injection achieves iron repletion in fewer doses (2) when compared with other available injectable iron formulations (5-6) available at NYU Langone Health, and thus may be useful to reduce travel burden and expedite full iron repletion in patients with iron deficiency. Iron-deficiency anemia is common in patients after placement of a ventricular assist device (VAD) for treatment of end-stage heart disease. This is a pilot study to test the feasibility of iron repletion with ferumoxytol injection in 20 eligible subjects with laboratory evidence of iron deficiency after placement of a VAD.

ELIGIBILITY:
Inclusion Criteria:

* Status post placement of durable ventricular assist device with stable clinical status for >30days
* Hemoglobin >6 g/dL AND <13 g/dL (men) or <12 g/dL (women) within last 90 days
* Serum ferritin <100 ng/mL OR Serum ferritin 100-299 ng/mL with transferrin saturation <20% within last 90 days
* Able and willing to provide written informed consent

Exclusion Criteria:

* Known hypersensitivity to Ferumoxytol injection or other intravenous iron preparation
* History of anaphylaxis
* Treatment with erythropoiesis stimulating agent or intravenous iron in last 3 months
* Renal failure on hemodialysis
* Respiratory failure on mechanical ventilation
* Disabling Stroke
* Ventricular assist device thrombosis
* Evidence of active gastrointestinal bleeding or other active blood loss
* Hospitalization <30 days
* Pregnant or breastfeeding women

Ages: 19 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Katz, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ferumoxytol Injection Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ferumoxytol Injection Treatment
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Successfully Complete Ferumoxytol Injection Treatment
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Ferumoxytol Injection Treatment
Number analyzed (Participants) | 1
percentage of participants | 100 (0)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Non-Systematic - subject reported and chart review
Arm/Group | Ferumoxytol Injection Treatment
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferumoxytol Injection Treatment (N=1)
Hospitalization - planned heart transplant, ICD and VAD removal (Surgical and medical procedures) | 1
Pneumoperitoneum (Injury, poisoning and procedural complications) | 1
Steriod Induced Hyperglycemia (Endocrine disorders) | 1
left shoulder disorder (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT04080908/Prot_SAP_000.pdf